CLINICAL TRIAL: NCT00002193
Title: A Randomized, Double-Blind, Placebo-Controlled Phase III Study to Evaluate the Safety and Efficacy of 141W94 Plus Current Nucleoside Therapy Versus Current Nucleoside Therapy Alone in Protease-Naive, HIV-Infected Children
Brief Title: Safety and Effectiveness of Giving Two Nucleoside Reverse Transcriptase Inhibitors Alone or in Combination With 141W94 to HIV-Infected Children Who Have Never Received Protease Inhibitors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Model: Parallel | Purpose: Treatment
Other Study IDs: 264C; PROA3004
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-06

CONDITIONS: HIV Infections
Keywords: HIV-1; Drug Therapy, Combination; HIV Protease Inhibitors; RNA, Viral; VX 478; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load
MeSH Terms: conditions — HIV Infections | interventions — amprenavir

INTERVENTIONS:
Drug: Amprenavir

SUMMARY:
The purpose of this study is to see if it is safe and effective to add a new protease inhibitor (PI), 141W94, to an anti-HIV regimen that includes 2 nucleoside reverse transcriptase inhibitors (NRTIs).

DETAILED DESCRIPTION:
In this double-blind, placebo-controlled, pediatric study, 210 patients are randomized to receive 2 NRTIs plus either 141W94 or placebo. Enrollment of patients is sequential: patients 13 to 18 years of age are enrolled first, followed by children < 13 when the appropriate pediatric dose has been determined. Patients who are unable to swallow capsules will be accrued when a liquid formulation becomes available.

ELIGIBILITY:
Inclusion Criteria

Your child may be eligible for this study if he/she:

* Is 6 months - 18 years of age.
* Is HIV-positive.
* Has a viral load (level of HIV in the body) greater than 10,000 copies/ml.
* Is able to take medications by mouth.
* Has consent of parent or legal guardian if under 18.
* Has a negative pregnancy test within 7 days of study entry.
* Agrees to practice abstinence or use effective methods of birth control for 1 month before and throughout the study.

Exclusion Criteria

Your child will not be eligible for this study if he/she:

* Has a serious illness, including any life-threatening infection or other chronic serious medical condition.
* Has an opportunistic (AIDS-related) infection or a serious bacterial infection.
* Is allergic to NRTIs.
* Is breast-feeding.
* Is unlikely to complete the study.
* Has received certain medications.
* Has received radiation therapy within the past 4 months, or will need to receive it during the study.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 210

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Children's Diagnostic Treatment Ctr, Fort Lauderdale, Florida
  - Saint Jude Children's Hosp / Dept of Infect Diseases, Memphis, Tennessee